CLINICAL TRIAL: NCT06452173
Title: Deep Learning-based Risk Prediction Model for Cerebrovascular Events in Patients With Carotid Artery Stenosis
Brief Title: Risk Prediction Model for Cerebrovascular Events in Carotid Artery Stenosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024-070-02; 2024-2-1072 (Other: Capitals Funds for Health Improvement and Research)
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Carotid Stenosis
Keywords: carotid stenosis; stroke; Risk prediction model; Deep-learning
MeSH Terms: conditions — Carotid Stenosis; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples Without DNA — blood and plaque specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high risk: Patients with cerebrovascular events within six months, including i. cerebral infarction in the middle cerebral artery territory on the side of carotid stenosis; ii. transient ischemic attack symptoms (including motor and sensory) in the hemisphere on the side of stenosis; and iii. transient amaurosis on the side of stenosis. This indicates an unstable condition and such patients are defined as high-risk carotid stenosis patients.
  Interventions: Diagnostic Test: Plasma; Diagnostic Test: carotid high-resolution magnetic resonance imaging
- low risk: Patients without cerebrovascular events within six months are defined as low-risk carotid stenosis patients.
  Interventions: Diagnostic Test: Plasma; Diagnostic Test: carotid high-resolution magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Plasma — Plasma levels of metabolites and some proteins will be further determined
Diagnostic Test: carotid high-resolution magnetic resonance imaging — Define plaque composition and morphological characteristics

SUMMARY:
Atherosclerotic carotid artery stenosis is a major cause of stroke, and early identification of high-risk patients combined with surgical intervention can significantly reduce stroke risk. Currently, stroke risk assessment in patients with carotid artery stenosis primarily relies on imaging indicators such as plaque morphology, composition, and degree of stenosis, with less emphasis on indicators directly related to inflammation, hemodynamics, and plaque instability. Certain circulating metabolites are closely linked to plaque progression and are direct risk factors for stroke. However, there is a lack of stroke risk prediction models for patients with carotid stenosis that incorporate these indicators, and the ability to identify high-risk patients needs improvement.

This study proposes using deep learning technology to integrate multidimensional data from plaque imaging, fluid dynamics, circulating metabolomics, and proteomics to construct an accurate prediction model for cerebrovascular events in patients with carotid artery stenosis. Additionally, it aims to explore markers of plaque instability characteristics based on plaque pathology. The study is expected to provide a basis for identifying high-risk patients with carotid artery stenosis, thereby laying the foundation for reducing stroke risk and improving long-term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with atherosclerotic carotid stenosis;
* Those who signed informed consent and volunteered to participate in this study.

Exclusion Criteria:

* Patients with combined severe stenosis of intracranial arteries;
* Patients with combined cardiogenic embolism, vasculitis, entrapment aneurysm and other related cerebral infarction;
* Combination of tumors, rheumatic immune system diseases, hematologic diseases and other diseases that change blood metabolism and proteomic characteristics;
* There are contraindications to magnetic resonance scanning and allergy to gadolinium contrast agent;
* Inability to cooperate in completing the relevant examinations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who met the enrollment criteria at Beijing Tiantan Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Cerebrovascular Events | Within six months from the date of consultation
  Patients will be categorized as having a cerebrovascular event if they meet one of the following indicators:
  i. cerebral infarction in the middle cerebral artery territory on the side of carotid stenosis; ii. transient ischemic attack symptoms (including motor and sensory) in the hemisphere on the side of stenosis; and iii. transient amaurosis on the side of stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, MD, Principal Investigator — Beijing Neurosurgical Institution
Locations (1):
- Beijing Tiantan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No